CLINICAL TRIAL: NCT06323590
Title: Refining the Role of Mid-induction Bone Marrow Biopsy in Acute Myeloid Leukemia: A Pilot
Brief Title: Refining the Role of Mid-induction Bone Marrow Biopsy in Acute Myeloid Leukemia: A Pilot Study
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Omer Jamy, Associate Professor, University of Alabama at Birmingham
Other Study IDs: UAB 2372; UAB (Other: UAB)
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort A: Patients with AML, receiving standard induction chemotherapy

SUMMARY:
The purpose of the study is to observe the outcomes of patients with acute myeloid leukemia who do not receive an immediate second round of chemotherapy after undergoing a standard mid-induction bone marrow biopsy.

DETAILED DESCRIPTION:
This will be a pilot study that will include patients with AML receiving intensive induction therapy with 7+3 +/- a third agent (for any actionable cytogenetics or mutations). All patients will have a planned mid-induction bone marrow assessment as standard of care. All patients will subsequently be observed for count recovery, regardless of bone marrow results and in the absence of peripheral blood disease proliferation, and an end of induction bone marrow biopsy will be performed either at count recovery or between days 28 and 42 in the absence of count recovery. Patients with complete remission (CR) will proceed to consolidation chemotherapy as determined by the treating investigator. Patients with refractory disease will proceed to further therapy as determined by the treating investigator. All patients will be followed for long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female, age ≥18
2. Patients with newly diagnosed AML (de novo or secondary), treated with intensive induction chemotherapy (7+3+/-3rd agent). The 3rd agent will be midostaurin for FLT3-mutant AML or gemtuzumab ozogamicin for core-binding factor AML. Patients on clinical trial with an investigational agent added to 7+3, may be enrolled on the protocol after discussion between the investigators and medical monitors.
3. Prior use of hypomethylating agents, lenalidomide, erythropoiesis stimulating agents and growth factors as allowed for treatment of myelodysplastic syndrome. Prior treatment for AML is not allowed.
4. Cardiac function: Ejection fraction >50-55%
5. Adequate organ function for receipt for induction chemotherapy
6. Patients with HIV and Hepatitis B or C should have controlled disease.
7. Females of childbearing potential must have a negative urine or serum pregnancy test prior to enrollment.

Exclusion Criteria:

1. Any other active malignancy requiring treatment or with expected survival ≤1 year.
2. Recipients of prior allogeneic stem cell transplant.
3. Patients with psychiatric illness or social situation that would limit compliance with the study requirements.
4. Patients with active CNS disease
5. Patients with APL
6. Received any investigational drugs within the 14 days prior to the first day of induction
7. Pregnant and/or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed AML (de novo or secondary), treated with intensive induction chemotherapy (7+3+/-3rd agent). The 3rd agent will be midostaurin for FLT3-mutant AML or gemtuzumab ozogamicin for core-binding factor AML.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
rates of complete remission | 28 days
  rates of complete remission in consecutive patients with AML, receiving standard induction chemotherapy, without intervening on the results of the mid-induction bone marrow biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Jamy, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States